CLINICAL TRIAL: NCT06307743
Title: A Multicenter, Open Label, Blind Endpoint, Clinical Trial to Evaluate the Efficacy and Safety of Rapid Local Ischemic Postconditioning in Acute Ischemic Stroke Patients Received Successful Thrombectomy Reperfusion
Brief Title: Rapid Local Ischemic Postconditioning in Acute Ischemic Stroke
Acronym: RAPID-SAVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Collaborators: Zhangzhou Municipal Hospital of Fujian Province (Other); Shanghai East Hospital (Other); First People's Hospital of Hangzhou (Other); RenJi Hospital (Other)
Responsible Party: Principal Investigator, Yueqi Zhu, Professor, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: RAPID-SAVE
Record Dates: First submitted 2024-03-04; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Acute Ischemic Stroke; Mechanical Thrombectomy; Ischemic Postconditioning; Brain Edema
MeSH Terms: conditions — Ischemic Stroke; Brain Edema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RL-IPostC 30 (Other): The RL-IPostC 30 protocol involved 5 cycles of blow block and restoration, each for 30 seconds.
  Interventions: Procedure: rapid local ischemic postconditioning
- RL-IPostC 60 (Other): The RL-IPostC 60 protocol involved 5 cycles of blow block and restoration, each for 60 seconds.
  Interventions: Procedure: rapid local ischemic postconditioning
- RL-IPostC 180 (Other): The RL-IPostC 180 protocol involved 5 cycles of blow block and restoration, each for 180 seconds.
  Interventions: Procedure: rapid local ischemic postconditioning

INTERVENTIONS:
Procedure: rapid local ischemic postconditioning — Rapid local ischemic postconditioning (RL-IPostC) is performed immediately (within 5 minutes) after revascularization. A balloon guiding catheter (BGC) positioned on ipsilateral C1 segment of internal carotid artery is inflated and deflated for the temporary occlusion of the antegrade flow.

SUMMARY:
The objective of this clinical trial is to determine whether rapid local ischemic postconditioning (RL-IPostC) is effective in preventing brain edema and safe in acute ischemic stroke (AIS) patients treated with mechanical thrombectomy. In this trial, researchers will block antegrade cerebral blood flow temporarily by the way of balloon inflation/deflation in AIS patients immediately after revascularization. It makes the ischemic reperfusion brain tissue have a capacity of adaptation through intermittent blood flow restoration. Researchers will evaluate the protective role and safety of different duration of balloon inflation/deflation. The optimal postconditioning intervention dose will be determined for further confirmative investigation.

DETAILED DESCRIPTION:
This will be an umbrella trial of testing the efficacy and safety of three postconditioning intervention doses. It will be a prospective, open-label, blinded endpoint, three-dose Bayesian Optimal Phase 2(BOP2) design trial with interim efficacy and safety monitoring. The maximum number of subjects for this trial is estimated as 135 patients. Eligible patients are 18 years or older with symptomatic large vessel occluded (LVO) AIS treated with mechanical thrombectomy (MT) achieving successful reperfusion defined as mTICI score 2b or 3. Patients will receive 5 cycles of balloon inflation/deflation at ipsilateral C1 segment of internal carotid artery (ICA) for the temporary occlusion of the restoration of antegrade blood flow. Three postconditioning intervention doses of 30s/30s, 60s/60s and 180s/180s were adopted for block and restore of blood blow. The primary outcome is a favorable binary outcome defined as no clinically meaningful brain swelling from baseline to 24 hours and no clinically meaningful infarction growth from baseline to 24 hours and no causally attributable serious adverse events (SAEs). It's a composite outcome of efficacy and safety outcome. Key secondary outcomes include efficacy outcome indicating no clinically meaningful brain swelling defined by cerebral spinal fluid (CSF) volume reduction≤5 mL from baseline to 24 hours and safety outcome indicating infarct volume growth>10 mL from baseline to 24 hours or causally attributable SAEs. Other secondary outcomes include change of brain net water uptake, midline shift and functional outcome. For each intervention dose, we will perform the interim analyses following pre-defined optimized Bayesian rule for early stopping to make a go/no-go decision when the number of enrolled patients reaches 10, 20, 30. The optimal intervention dose will be determined according to the number of patients reach the primary endpoints in different groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Presenting with symptoms consistent with acute ischemic stroke
3. Pre-stroke mRS score 0-1
4. Baseline NIHSS score≥6
5. Endovascular treatment can be initiated (femoral puncture) within 24 hours from stroke onset (stroke onset time is defined as last known well time)
6. Occlusion of the intracranial internal carotid artery, or the middle cerebral artery(M1 or M2) confirmed by CTA or MRA, and is the culprit artery
7. Alberta Stroke Program Early CT Score (ASPECTS) (based on non-contrast CT) >5 on noncontrast computed tomography (NCCT) for stroke onset time less than 6 hours, infarct Core < 70 ml (defined as rCBF <30% on CT perfusion) and mismatch ratio > 1.2 (penumbra defined as Tmax >6 seconds volume) for stroke onset time between 6 and 24 hours.
8. Embolism verified as the etiology of occluded artery and mTICI 2b or 3 regained after mechanical thrombectomy
9. Informed consent signed

Exclusion Criteria:

1. Stenosis of the proximal middle cerebral artery, internal carotid artery, or common carotid artery (≥50%) of the culprit artery
2. Multiple vascular embolism on different pathways (not refers to the ipsilateral middle artery and anterior artery)
3. Pre ischemic stroke or transient ischemic attack within past 3 months
4. The expected survival time is less than 6 months, could not be followed at 90 days (such as patient with malignant tumor)
5. Currently pregnant, mental disease, advanced hepatic and renal insufficiency, severe heart failure
6. Participation in other interventional randomized clinical trials that may confound the outcome assessment of the trial
7. Other circumstances that the investigator considers inappropriate for this trial

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants without clinically meaningful cerebral swelling, significant increase in infarct volume from baseline and intervention-related serious adverse events. | 24 hours after procedure
  No clinically meaningful cerebral swelling defined as volume reduction of cerebrospinal fluid ≤ 5 mL from baseline. No significant increase in infarct volume from baseline defined as an increase in infarct volume of ≤ 10 mL. Intervention-related serious adverse events defined as SAEs specifically related to RL-IPostC other than mechanical thrombectomy.

SECONDARY OUTCOMES:
Rate of participants without clinically meaningful cerebral swelling | 24 hours after procedure
  No clinically meaningful brain swelling defined by CSF volume reduction≤5 mL from baseline to 24 hours.
Rate of participants with significant increase in infarct volume from baseline or intervention-related serious adverse events. | 24 hours after procedure
  Significant increase in infarct volume from baseline defined as an increase in infarct volume of more than 10 mL. Intervention-related serious adverse events defined as SAEs specifically related to RL-IPostC other than mechanical thrombectomy.
Change in volume of cerebrospinal fluid (∆CSF72) at 72 hours | 72 hours after procedure
  Change in volume of cerebrospinal fluid (∆CSF72) at 72 hours from baseline
Change of net water uptake (∆NWU24) at 24 hours | 24 hours after procedure
  Change of net water uptake (∆NWU24) at 24 hours from baseline
Change of net water uptake (∆NWU72) at 72 hours | 72 hours after procedure
  Change of net water uptake (∆NWU72) at 72 hours from baseline
Midline shift at 24 hours | 24 hours after procedure
  Distance of midline shift at 24 hours (in millimeters at the level of the septum pellucidum)
Midline shift at 72 hours | 72 hours after procedure
  Distance of midline shift at 72 hours (in millimeters at the level of the septum pellucidum)
Change of NIHSS at 24 hours | 24 hours after procedure
  Change of NIHSS at 24 hours from baseline
Early therapeutic response to treatment | 24 hours after procedure
  Decrease in the NIHSS score of ≥8 from baseline or an NIHSS score of 0 to 2 at 24 hours)
Good outcome at 90 days | 90 days after procedure
  Proportion of mRS score of 0 to 2 at 90 days
Excellent outcome at 90 days | 90 days after procedure
  Proportion of mRS score of 0 to 1 at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Yueqi Zhu, MD, Principal Investigator — Shanghai Jiao Tong University Affiliated Sixth People's Hospital

IPD SHARING:
Plan to Share IPD: No